CLINICAL TRIAL: NCT06168058
Title: Randomized Controlled, Single-Blinded, Parallel-Group Trial of Ovarian Vein and Pelvic Vein Embolization in Women With Chronic Pelvic Pain and Pelvic Varices (EMBOLIZE) Trial
Brief Title: Trial of Ovarian Vein and Pelvic Vein Embolization in Women With Chronic Pelvic Pain and Pelvic Varices
Acronym: EMBOLIZE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Society of Interventional Radiology Foundation (Other); VIVA Physicians (Other); Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-08026405
Record Dates: First submitted 2023-11-14; First posted 2023-12-13 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pelvic Pain Syndrome; Pelvic Pain; Pelvic Varices; Pelvic Congestive Syndrome; Pelvic Pain Syndrome
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Transcatheter Venography (Sham Comparator)
  Interventions: Diagnostic Test: Transcatheter Venography
- Bilateral Ovarian Vein Embolization (Experimental): Transcatheter Venography plus Bilateral Ovarian Vein Embolization.
  Interventions: Diagnostic Test: Transcatheter Venography; Procedure: Bilateral ovarian vein embolization

INTERVENTIONS:
Diagnostic Test: Transcatheter Venography — Venographic assessment of ovarian veins and internal iliac veins
  Other Names: Diagnostic Venography
Procedure: Bilateral ovarian vein embolization — Intervention will include sclerosis of pelvic varices and coil embolization of the bilateral ovarian veins.
  Other Names: Ovarian vein and pelvic vein embolization
  Arms: Bilateral Ovarian Vein Embolization

SUMMARY:
The purpose of this study is to see if a randomized controlled trial of ovarian vein and pelvic vein embolization versus venography alone could determine outcomes for women with chronic pelvic pain and pelvic varicose veins.

The data gathered will assist in addressing changes in quality of life in patients who have ovarian/pelvic vein embolization versus no embolization.

DETAILED DESCRIPTION:
The study is a randomized research trial of bilateral ovarian vein embolization (OVE) and pelvic vein embolization (PVE) in women with chronic pelvic pain (CPP), dilated and incompetent ovarian veins ≥6mm and pelvic varices (≥1 veins, >5 mm diameter) to assess for change in pain. Pain will be assessed by visual analog scale (VAS) and other relevant, validated quality of life metrics including the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v.1.0 - Pain Intensity, Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v1.2 - Global Health, Patient Global Impression of Change (PGIC) and EuroQol five-dimension (EQ 5D). The target population includes women age greater than or equal to 18 years who are pre-menopausal and have symptoms, and clinical and imaging findings corresponding to Pelvic Venous Disease (PeVD). Subjects will be randomized in a 1:1 fashion to embolization (treatment group) or venography only (control group). Follow-up will be assessed weekly and at 1, and 3 months and 6 months post procedure to assess for changes in quality of life in patients who receive ovarian/pelvic vein embolization versus no embolization.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of venous origin chronic pelvic pain for greater than 6 months (VAS ≥7 as determined by 4 consecutive weeks of baseline self-assessments) despite non-vascular therapy as delineated by the following criteria:

   * Pain exacerbated by walking, standing or lifting
   * Symptoms are at least partially alleviated by lying down
   * Prolonged post-coital ache
   * Absence of non-venous origin CPP as determined by Gynecology examination
2. Symptoms-Varices-Pathophysiology Classification18 including of one of the following:

   •S2V2PBGV,R,NT, S2V2PRGV,R,NT , S2V2PLGV,R,NT, with or without S2V2 PBIIV,R,NT, S2V2 PLIIV,R,NT, S2V2 PRIIV,R,NT
3. CT, TAUS and diagnostic venography (if needed) imaging review for pelvic venous imaging factors

   * Left or right ovarian vein diameter greater than or equal to 6 mm as documented by TAUS or CT
   * Presence of intrabdominal/pelvic varices as documented by TAUS or CT (≥1 veins, >5 mm diameter)
   * Presence of venous reflux in ovarian and/or internal iliac veins without evidence of hemodynamically significant stenosis

Exclusion Criteria:

* Female <18 years of age
* Pregnancy (positive pregnancy test)
* Female subject who plans to become pregnant during study period
* Female subject who is actively breastfeeding
* Patient who is post-menopausal or anovulatory with hormone suppression
* History of prior hysterectomy
* Prior ovarian vein embolization or ovarian vein ligation
* Inability to tolerate endovascular procedure due to acute illness or general health
* Planned simultaneous treatment with nerve blocks during the duration of the study
* Laparoscopy or planned surgical intervention during the duration of the study
* Known allergy to sclerosant, coil, stent or catheter components including nickel allergy
* Any iliac vein stenosis determined identified by the investigator on pelvic DUS, CT venogram, and/or Catheter Venography and deemed significant for exclusion by study patient review committee.
* Any renal vein stenosis with resultant renal hilar varices/collaterals and lumbar collaterals identified by the investigator on pelvic DUS, CT venogram, and/or Diagnostic Venography and deemed significant for exclusion by study patient review committee.
* Presence of isolated extra-pelvic vulvar and/or lower extremity varices without intrabdominal pelvic varices. Primary S3 categorization study exclusion.
* Serious medical conditions that might preclude full participation in the study to the desired endpoint (e.g., uncontrolled diabetes, malignancy, COPD, MI, CHF, etc.)
* Severe allergy to iodinated or gadolinium-based contrast refractory to steroid premedication
* Severe renal impairment (on chronic dialysis or estimated GFR <30 mL/min)
* Hemoglobin <8.0 g/dL, uncorrectable INR >3.0 or platelet count <75,000/microliter
* Inability to provide informed consent or to comply with study assessments
* Post thrombotic IVC, iliac or ovarian vein changes

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) for pelvic pain | Weekly for 4 weeks prior to Day 1 and at 30, 90 and 180 day follow up
  The VAS pain score is a standard scale from 0 to 10, defining 0 as ''no pain'' and 10 ''worst pain possible.''

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) 3A Pain Intensity Scale | Weekly for 4 weeks prior to Day 1 and at 30, 90 and 180 day follow up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) 3A Pain Intensity Scale assess how much a person hurts. The scale ranges from 1-5, defining 1 as ''no pain'' and 5 ''very severe pain.''
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) 10 Pain Intensity Scale | Weekly for 4 weeks prior to Day 1 and at 30, 90 and 180 day follow up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health measures assess an individual's physical, mental, and social health. The scale scores from from 5 to 1 with 5 = "Excellent" and 1= "Poor ".
Change in Patient Global Impression of Change (PGIC) | 30, 90 and 180 day follow up
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale with 1= "Very Much Improved" and 7= "Very Much Worse".
Change in EuroQol five-dimension (EQ-5D) scale | Weekly for 4 weeks prior to Day 1. Then at 30, 90 and 180 day follow up
  The EuroQol five-dimension (EQ-5D) is a concise, generic measure of self-reported health at each visit. Patients will tick the one box that best describes their health on that day. This scale will measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.The scale is numbered from 0 to 100. =100 means the best health the patient can imagine and 0 means the worst health the patient can imagine,.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald S Winokur, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Weill Cornell Medicine, New York, New York
  - UNC School of Medicine, Chapel Hill, North Carolina
  - Lake Washington Vascular, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No